CLINICAL TRIAL: NCT06287281
Title: Repercussions on Spinal Posture Before and After Wearing High-heeled Shoes in a Sample of Young Women: Cross-sectional Pilot Study
Brief Title: High-heeled Shoes in a Sample of Young Women
Status: Recruiting | Type: Observational
Sponsor: Manusapiens (Other)
Responsible Party: Sponsor
Other Study IDs: Heel01
Record Dates: First submitted 2024-02-11; First posted 2024-03-01 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Low Back Pain; Healthy
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: heel hight shoes — stand upright for 2 hours wearing your own shoes with heels at least 7 cm high

SUMMARY:
At a postural level, many doctors, physiotherapists and chiropractors are convinced that lower back pain induced by heels is due to an increase in lumbar lordosis associated with an anterior pelvic tilt; this thought is even shared by the American Chiropractic Association and the American Physical Therapy Association.

Furthermore, in most of the websites consulted, even by non-experts, the reason for the onset of spinal pain is attributed to hyperlordosis and pelvic anteversion. However, this thought is not entirely in agreement with other scientific publications. Therefore it is necessary to pay attention to online searches which often answer these questions without taking EBM into account.

None of the studies reported above take into consideration the time factor. In fact, all the studies have evaluated the immediate changes brought about by heel raising. Women who complain of lower back pain when wearing high-heeled shoes rarely experience pain as soon as they start wearing them.

The objective of the research arises from these considerations. The aim of this study (primary outcome) is to investigate whether wearing high-heeled shoes for at least 2 hours modifies the spinopelvic parameters compared to the barefoot condition and as soon as the shoes are worn.

The secondary outcome will be to verify in the sample analyzed whether there are different behaviors between the subgroups of those who have complained in their anamnesis and those who have never complained of lower back pain when using high-heeled shoes for a few hours.

DETAILED DESCRIPTION:
A three-dimensional analysis of the posterior surface will be performed with the Formetric 4D® rasterstereographic device (Diers International GmbH, Schlangenbad, Germany).

Participants will be given a questionnaire which investigates:

* Age, weight, height of the participants;
* Any pain in the spine (measured by NPS) usually reported by subjects after using high-heeled shoes;
* Type of profession;
* Frequency with which the subjects wear the heeled shoe (how many hours per week);
* Heel height of the shoe with which they participate in the clinical study;
* Any spinal pain (measured by NPS) after wearing heeled footwear for the study period.

This last data will be filled in at the end of the evaluation.

For the evaluation of the secondary outcome, on the basis of the data from the medical history sheet, the sample will be divided into two groups:

1. The first group (group A, ASYMPTOMATIC) includes subjects who during daily life do not report spinal pain after wearing high-heeled shoes;
2. The second group (group S, SYMPTOMATIC) is made up of participants who usually complain of more or less intense pain after using the shoe.

The subjects will be asked to bring their own pair of shoes with a heel that is at least 8.7 cm, the average height reported by the work of Schroeder and Hollander, where average height means the difference between the height of the heel and the height of the raised part at the forefoot level (plateau). A particular heel width will not be required, because it seems that the height of the heel influences muscle activation, in particular the paravertebral muscles, while the width of the heel has no significant effects on them.

Conversely, amplitude has a greater influence on balance when standing and while walking.

Three evaluation will be performed:

1. first evaluation in neutral position with bare feet (T0)
2. second evaluation in neutral position wearing shoes (T1);
3. third evaluation like the previous one but at least 2 hours apart, in which it will be required to remain standing still or walk (T2).

Statistic analysis

A descriptive analysis of the population will be performed to determine the mean values and standard deviations (SD) of both the combined group and the subgroups A and S. T-tests for independent data will be used to verify whether there are any significant differences between the two subgroups .

The distribution of the data will be verified using graphical representation. If the distribution is normal (p <0.05) for the comparison between T1 vs T2 the t-test for paired data will be used and between the subgroups (T1S vs T1A and T2S vs T2A) t-test for independent data with statistical significance accepted for p values <0.05. ANOVA will be used to simultaneously compare the pre and post of both groups.

If the data does not have a normal distribution (p >0.05) the Wilcoxon test will be used for the comparison between the T1 vs T2 data of the total group and the Mann-Whitney U test for the comparison between subgroups (T1S vs T1A and T2S vs T2A). The Friedman test will be used to simultaneously compare the pre and post of both groups.

ELIGIBILITY:
Inclusion Criteria:

* female subjects aged between 20 and 40 years
* Usual users of shoes with heels at least 7 cm high, with a frequency of at least twice a week and/or less than 3 hours/week

Exclusion Criteria:

* structural or neurological anomalies that may prevent you from remaining weight-bearing, for approximately 2 hours, with shoes having a heel (difference between the heel and the plateau) of at least 7 cm high;

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Usual female users of shoes with heels at least 7 cm high, with a frequency of at least twice a week and/or less than 3 hours/week
Sampling Method: Non-Probability Sample
Enrollment: 34 (Estimated)
Dates: Start 2023-12-15 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
effect of high-heeled shoes on trunk inclination | 2 hours after wearing high heels
  The aim of this study is to investigate whether wearing high-heeled shoes for at least 2 hours modifies the flexion of the antero-posterior trunk (measured as the angle between the vertical and the line that passes through the prominent cervical vertebra and the line that connects the two dimples) compared to the barefoot condition and as soon as the shoes are worn.
effect of high-heeled shoes on pelvic inclination | 2 hours after wearing high heels
  The aim of this study is to investigate whether wearing high-heeled shoes for at least 2 hours modifies the pelvic inclination angle (the angle between the vertical and the tangent to the lumbosacral junction) compared to the barefoot condition and as soon as the shoes are worn.
effect of high-heeled shoes on lordotic angle | 2 hours after wearing high heels
  The aim of this study is to investigate whether wearing high-heeled shoes for at least 2 hours modifies the lordotic angle (angle measured between the tangents of the thoracolumbar junction and the lumbosacral junction) compared to the barefoot condition and as soon as the shoes are worn.
effect of high-heeled shoes on kyphotic angle | 2 hours after wearing high heels
  The aim of this study is to investigate whether wearing high-heeled shoes for at least 2 hours modifies the kyphotic angle (angle measured between the tangents of the cervicothoracic junction and the thoracolumbar junction) compared to the barefoot condition and as soon as the shoes are worn.
effect of high-heeled shoes on lumbar arrow | 2 hours after wearing high heels
  The aim of this study is to investigate whether wearing high-heeled shoes for at least 2 hours modifies the lumbar arrow (horizontal distance in millimeters of the lumbar spine from the virtual vertical line that passes through the kyphotic apex) compared to the barefoot condition and as soon as the shoes are worn.
effect of high-heeled shoes on cervical arrow | 2 hours after wearing high heels
  The aim of this study is to investigate whether wearing high-heeled shoes for at least 2 hours modifies the cervical arrow (horizontal distance in millimeters of the cervical spine from the virtual vertical line that passes through the kyphotic apex) compared to the barefoot condition and as soon as the shoes are worn.

SECONDARY OUTCOMES:
different response on trunk inclination between the subgroups (suffering from back pain and asymptomatic) | 2 hours after wearing high heels
  The secondary outcome will be to verify in the sample analyzed whether there are different behaviors of the flexion of the antero-posterior trunk (measured as the angle between the vertical and the line that passes through the prominent cervical vertebra and the line that connects the two dimples) between the subgroups of those who suffer from low-back pain and those who have never complained of low-back pain when using high-heeled shoes for a few hours.
different response on pelvic inclination between the subgroups (suffering from back pain and asymptomatic) | 2 hours after wearing high heels
  The secondary outcome will be to verify in the sample analyzed whether there are different behaviors of the pelvic inclination angle (the angle between the vertical and the tangent to the lumbosacral junction) between the subgroups of those who suffer from low-back pain and those who have never complained of low-back pain when using high-heeled shoes for a few hours.
different response on lordotic angle between the subgroups (suffering from back pain and asymptomatic) | 2 hours after wearing high heels
  The secondary outcome will be to verify in the sample analyzed whether there are different behaviors of the lordotic angle (angle measured between the tangents of the thoracolumbar junction and the lumbosacral junction) between the subgroups of those who suffer from low-back pain and those who have never complained of low-back pain when using high-heeled shoes for a few hours.
different response on kyphotic angle between the subgroups (suffering from back pain and asymptomatic) | 2 hours after wearing high heels
  The secondary outcome will be to verify in the sample analyzed whether there are different behaviors of the kyphotic angle (angle measured between the tangents of the cervicothoracic junction and the thoracolumbar junction) between the subgroups of those who suffer from low-back pain and those who have never complained of low-back pain when using high-heeled shoes for a few hours.
different response on lumbar arrow between the subgroups (suffering from back pain and asymptomatic) | 2 hours after wearing high heels
  The secondary outcome will be to verify in the sample analyzed whether there are different behaviors of the lumbar arrow (horizontal distance in millimeters of the lumbar spine from the virtual vertical line that passes through the kyphotic apex) between the subgroups of those who suffer from low-back pain and those who have never complained of low-back pain when using high-heeled shoes for a few hours.
different response on cervical arrow between the subgroups (suffering from back pain and asymptomatic) | 2 hours after wearing high heels
  The secondary outcome will be to verify in the sample analyzed whether there are different behaviors of the cervical arrow (horizontal distance in millimeters of the cervical spine from the virtual vertical line that passes through the kyphotic apex) between the subgroups of those who suffer from low-back pain and those who have never complained of low-back pain when using high-heeled shoes for a few hours.

CONTACTS AND LOCATIONS:
Overall Officials: Saverio Colonna, MD, Principal Investigator — Spine Center
Locations (1):
- Spine Center, Bologna, Italy

REFERENCES:
- [Background] Lee CM, Jeong EH, Freivalds A (2001) Biomechanical effects of wearing high-heeled shoes. Int J Indust Ergonom 28:321-326
- [Background] de Oliveira Pezzan PA, Joao SM, Ribeiro AP, Manfio EF. Postural assessment of lumbar lordosis and pelvic alignment angles in adolescent users and nonusers of high-heeled shoes. J Manipulative Physiol Ther. 2011 Nov;34(9):614-21. doi: 10.1016/j.jmpt.2011.09.006. PMID 22078999
- [Background] Dai M, Li X, Zhou X, Hu Y, Luo Q, Zhou S. High-heeled-related alterations in the static sagittal profile of the spino-pelvic structure in young women. Eur Spine J. 2015 Jun;24(6):1274-81. doi: 10.1007/s00586-015-3857-6. Epub 2015 Mar 10. PMID 25753007
- [Background] de Lateur BJ, Giaconi RM, Questad K, Ko M, Lehmann JF. Footwear and posture. Compensatory strategies for heel height. Am J Phys Med Rehabil. 1991 Oct;70(5):246-54. PMID 1910649
- [Background] Franklin ME, Chenier TC, Brauninger L, Cook H, Harris S. Effect of positive heel inclination on posture. J Orthop Sports Phys Ther. 1995 Feb;21(2):94-9. doi: 10.2519/jospt.1995.21.2.94. PMID 7711763
- [Background] Schroder G, Kundt G, Otte M, Wendig D, Schober HC. Impact of pregnancy on back pain and body posture in women. J Phys Ther Sci. 2016 Apr;28(4):1199-207. doi: 10.1589/jpts.28.1199. Epub 2016 Apr 28. PMID 27190453
- [Background] Gerber SB, Costa RV, Grecco LA, Pasini H, Marconi NF, Oliveira CS. Interference of high-heeled shoes in static balance among young women. Hum Mov Sci. 2012 Oct;31(5):1247-52. doi: 10.1016/j.humov.2012.02.005. Epub 2012 Jun 27. PMID 22742722
- [Background] Han D. Muscle activation of paraspinal muscles in different types of high heels during standing. J Phys Ther Sci. 2015 Jan;27(1):67-9. doi: 10.1589/jpts.27.67. Epub 2015 Jan 9. PMID 25642040
- [Background] Russell BS. The effect of high-heeled shoes on lumbar lordosis: a narrative review and discussion of the disconnect between Internet content and peer-reviewed literature. J Chiropr Med. 2010 Dec;9(4):166-73. doi: 10.1016/j.jcm.2010.07.003. Epub 2010 Oct 14. PMID 22027108
- [Background] Kwon YJ, Song M, Baek IH, Lee T. The effect of simulating a leg-length discrepancy on pelvic position and spinal posture. J Phys Ther Sci. 2015 Mar;27(3):689-91. doi: 10.1589/jpts.27.689. Epub 2015 Mar 31. PMID 25931709

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-10): https://cdn.clinicaltrials.gov/large-docs/81/NCT06287281/Prot_SAP_000.pdf